CLINICAL TRIAL: NCT05468177
Title: A Multiple-Center,Single-arm Clinical Study of Cetuximab in Combination With Anti-PD-1 and mFOLFOX Treat For RAS/BRAF wt Locally Advanced or Metastatic Right-Sided Colon Cancer
Brief Title: Cetuximab in Combination With Anti-PD-1 and mFOLFOX Treat For RAS/BRAF wt Right-Sided Colon Cancer
Acronym: CIFOXRC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Collaborators: Huangshi Central Hospital (Other); Central Hospital of Xiaogan (Other); Ezhou Central Hospital (Unknown); Jingzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB20220165
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-01

CONDITIONS: Colonic Neoplasms
Keywords: neoadjuvant chemotherapy; cetuximab; right colon cancer; immunotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neoadjuvant chemotherapy (Experimental): Cetuximab+ mFOLFOX+ Anti-PD-1+Surgery
  Interventions: Combination Product: neoadjuvant chemotherapy

INTERVENTIONS:
Combination Product: neoadjuvant chemotherapy — Cetuximab: 500mg/m2,day1, every 2 weeks. mFOLFOX: oxaliplatin 85mg/m2, day 1;LV 400mg/m2, day 1;5-FU 400mg/m2, day 1, then 1200mg/ (m2•d) ×2days(total 2400mg/m2, infusion 46-48h) (every 2 weeks).
  Anti-PD-1(Sintilimab Injection):200mg every 3 weeks. Surgery will be performed after 4 cycles for locally advanced or initially resectable metastatic right colon cancer.If the initial unresectable metastatic right colon cancer were converted into resectable metastases, and surgery will be performed. Patients who failed to convert after 6 cycles of treatment will be withdrawn from the study.Cetuximab +mFOLFOX was treat for 8 cycles, and Anti-PD-1 was treated for one year in the perioperation period unless disease progression, toxicity intolerance, initiation of new anti-tumor therapy.

SUMMARY:
We plan to evaluate the efficacy and safety of cetuximab combined with anti-PD-1 and mFOLFOX6 in the treatment of RAS/BRAF WT locally advanced or metastatic right colon cancer

DETAILED DESCRIPTION:
According to the World Health Organization, colorectal cancer (CRC) is the third most common cancer in men and the second most common cancer in women worldwide. CRC is estimated to kill 551,269 patients worldwide each year, accounting for 5.8% of cancer deaths.Despite recent development in treatment, locally advanced or metastatic colon cancer (CC) represents a major therapeutic challenge. Presently, the standard therapeutic approach for CC is surgery and/or adjuvant chemotherapy. Nevertheless,several studies showed that neoadjuvant chemotherapy (NAC) is a more effective treatment option.Immune checkpoint inhibition (ICI) directed against programmed death-1 (PD-1) is highly effective and has become the standard of care for patients with dMMR metastatic colorectal cancers (mCRCs). In contrast, the same regimens have shown poor response rates in patients with pMMR mCRCs.Due to the high ORR rate of cetuximab combined with chemotherapy and the microenvironment with high immune infiltration of right colon cancer, it may be more sensitive to ICI.

This study consisted of two phases: phase I consisted of 25 patients; if > 11 patients responded, the trial will continue to phase II, and a total of 66 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. RAS and BARF wild-type right colon adenocarcinoma (cecum, ascending colon, transverse colon excluding splenic flexure) confirmed by histopathology;
2. Locally advanced right colon cancer should be assessed as T3 (invading muscularis propria ≥5mm) or T4 according to abdominal CT;
3. Metastatic right colon cancer should conforms to the definition of oligometastasis of colorectal cancer in ESMO guidelines: the number of organs involved is ≤2 (occasionally 3), and the number of metastases is usually ≤5 or occasionally more.
4. At least one measurable lesion according to RECIST1.1;
5. ECOG score 0-1;
6. The expected survival time is more than 3 months;
7. Adequate organ function: total bilirubin ≤1.5 x upper limit of normal (ULN) , aspartate aminotransferase and alanine aminotransferase ≤2.5 x ULN (if patient with liver metastasis, total bilirubin ≤3 x ULN, aminotransferase and alanine aminotransferase ≤5x ULN) ,alkaline phosphatase ≤2.5 x ULN (if liver metastases≤5x ULN, if bone metastases ≤10 x ULN);LDH < 1500 U/L;Serum creatinine≤1.5 x ULN l or creatinine clearance rate ≤ 60 mL /min;ANC≥1.5×109 /L, platelet count ≥75×109 /L, Hb ≥90 g/L, WBC ≥3.0×109 /L;
8. Capable of providing informed consent, or if not capable, a legally authorized representative is capable of providing informed consent.

Exclusion Criteria:

* 1.Early stage right colon cancer. 2. Received chemotherapy or biotherapy in the past . 3. uncontrollable infection, or received antibiotic treatment within 72 hours prior to receive chemotherapy; 4. Myelodysplastic syndrome or other hematopoietic abnormalities; 5. Other malignant tumors (except carcinoma in situ and basal cell carcinoma) during this year; 6. Patients with central nervous system metastasis; 7.≥ CTCAE Grade 2 unrecovered AEs due to prior treatment (excluding anemia, hair loss, skin pigmentation).Patients with unrecovered neurotoxicity ≥ CTCAE grade 3 due to platinum-based drugs.

  8. Other diseases, such as active tuberculosis, infect HIV, AIDS, hepatitis B (patient withHBV-DNA <500IU/ml,and normal liver function can be included), positive test for hepatitis C virus, uncorrectable electrolyte disorder;ascites, pleural effusion or hydropericardium that required drainage in the past 4 weeks.With intestinal obstruction, gastrointestinal bleeding, pulmonary fibrosis or interstitial pneumonia, renal failure, hepatic failure , or cerebrovascular disease.

  9. Uncontrolled diabetes was defined as HbA1c >7.5% after the use of antidiabetic drugs, or uncontrolled hypertension was defined as systolic/diastolic blood pressure >140/90 mmHg after the use of antihypertensive drugs.

  10. Myocardial infarction,severe/unstable angina, NYHA III or IV congestive heart failure within the past 12 months.

  11. Patients who are allergic to the therapeutic drugs in this study; 12. With mental or nervous system diseases who are unable to cooperate; 13. Pregnant or lactating women;Childbearing age women refuse to accept contraceptive measures; 14.Active autoimmune disease, a history of autoimmune disease, accepting corticosteroid or immunosuppressants, or accepting hormone replacement therapy (such as thyroxine, insulin, etc).

  15. Received live vaccine within 30 days (seasonal influenza vaccine is allowed because it is inactivated) 16.Treated with any other investigational drug or participated in another interventional clinical trial within 30 days of the screening period; undergo surgery within 30 days (except for diagnostic biopsy, surgical incision should be completely healed prior to administration of the study drug).Received radiation therapy within 30 days.

  17. Other serious medical conditions made the investigator consider the patients ineligible for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | an average of 6 to 12 weeks after surgery
  percentage of patients showing complete response (CR) or partial response (PR) as best response according to RECIST1.1

SECONDARY OUTCOMES:
disease free survival (DFS) | UP to 3 years
  DFS is defined as the time from treatment initiation to the date of first documentation of disease recurrence or death due to any cause
R0 resection rate | an average of 6 to 12 weeks after surgery
  The percentage of patients whose post-operative pathology indicate negative margin is observed under microscope

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No